CLINICAL TRIAL: NCT06295770
Title: A Single-Center Phase 2 Open-Label Trial Evaluating the Efficacy and Safety of Obinutuzumab in Treatment of Fibrillary Glomerulonephritis
Brief Title: Obinutuzumab in Treatment of Fibrillary Glomerulonephritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ladan Zand, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-006712
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Fibrillary Glomerulonephritis
MeSH Terms: interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Obinutuzumab in Treatment of Fibrillary Glomerulonephritis (Experimental): Patients with biopsy proven fibrillary GN who have >1 gram/24 hour of proteinuria and eGFR ≥ 20 ml/min/BSA will be treated with Obinutuzumab.
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab 1g IV on day one and 1 g IV on day 15, followed by identical course at month 6.
  Other Names: Gazyva

SUMMARY:
The purpose of this research is to learn if Obinutuzumab is effective and safe in treating patients with fibrillary glomerulonephritis (FGN).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Biopsy proven fibrillary glomerulonephritis
* Proteinuria > 1.0 g/24hrs prior to initiation of immunosuppressive therapy
* eGFR ≥ 20 ml/min/BSA

Exclusion Criteria:

* Secondary FGN (due to monoclonal gammopathy, autoimmune disease or malignancy)
* Presence of a secondary pathology on biopsy (e.g. diabetic nephropathy)
* Hepatitis B, C or HIV positive
* Pregnant or breast-feeding
* Active infection
* Kidney transplant
* Anemia with Hgb < 8.0 g/dL
* Thrombocytopenia with platelet count < 100'000
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complication
* Patients who have received cyclophosphamide in the last 6 months
* Patients who have received ACTH and/or mycophenolate mofetil in the last 30 days
* Patient who are on prednisone therapy at a dose > 10 mg/day in the last 15 days
* Patients who received rituximab previously with CD20 count of < 5 cells/microliter at the time of enrollment
* For women who are not postmenopausal (greater than or equal to [>/=] 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of less than (<) 1 percent (%) per year, during the treatment period and for at least 18 months after the last dose of study drug
* For men: agreement to remain abstinent or use two adequate methods for contraception, including at least one method with failure rate of less than 1% per year during the treatment period and for at least 6 months (180 days) after the last dose of drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in proteinuria from baseline to 12 months post treatment with Obinutuzumab | Baseline, 6 months, 12 months
  Measured using 24-hour urine collection reported in mg/24h

SECONDARY OUTCOMES:
Change in proteinuria from baseline to 6 months post treatment with Obinutuzumab | Baseline, 6 months
  Measured using 24-hour urine collection reported in mg/24h
Rate of complete or partial remission | 6 months, 12 months
  Complete remission: Proteinuria < 0.5g/24 hrs. and no more than 20% decline in eGFR Partial remission: 50% reduction in proteinuria and proteinuria < 3.5 g/24hrs and no more than 20% decline in eGFR
Improvement in serum albumin | Baseline, 6 months, 12 months
  Blood serum collected and reported in g/dL
Stabilization of kidney function | Baseline, 6 months, 12 months
  Stabilization is defined as no more than 20% decline in eGFR at 6 months and 12 months. Blood serum collected and reported in mL/min/BSA.
Serious Adverse Events (SAEs) | Day 1-12 months
  Rate of all Serious Adverse Events (SAEs) including serious infection defined as severe UTI or pyelonephritis, pneumonias or other systemic infections requiring hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Ladan Zand, Principal Investigator — Mayo Clinic; Fernando Fervenza, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No